CLINICAL TRIAL: NCT00932607
Title: SUBLIVAC® Birch Prospective, Randomized, Open, Blinded Endpoint (PROBE) Study
Brief Title: SUBLIVAC® Birch PROBE Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SB/0027
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Seasonal Rhinitis and/or Rhinoconjunctivitis; Birch Pollen Allergy
Keywords: seasonal; rhinitis; rhinoconjunctivitis; birch pollen; immunotherapy; sublingual
MeSH Terms: conditions — Rhinitis | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Staloral Birch (Active Comparator): Start with 1 puff of Staloral Birch 10 I.R./ml on day one, 2 puffs on day two and increase by 2 puffs until at day six 10 puffs are reached. At day seven 1 puff of Staloral Birch 300 I.R./ml is taken, at day eight 2 puffs and day nine 4 puffs. From then on 4 puffs daily are taken.
  Duration of treatment: 16-20 weeks per subject (at least 12 weeks for subjects with hazel or alder allergy).
  Interventions: Drug: sublingual immunotherapy
- SUBLIVAC Birch (Experimental): Start with 1 drop daily of SUBLIVAC Birch and increase by 1 drop daily, until the maintenance dose of 5 drops is reached. This maintenance dose should then be taken daily.
  Duration of treatment: 16-20 weeks per subject (at least 12 weeks for subjects with hazel or alder allergy).
  Interventions: Drug: sublingual immunotherapy

INTERVENTIONS:
Drug: sublingual immunotherapy — Start with 1 drop daily of SUBLIVAC Birch and increase by 1 drop daily, until the maintenance dose of 5 drops is reached. This maintenance dose should then be taken daily. Or 1 puff of Staloral Birch 10 I.R./ml on day one, 2 puffs on day two and increase by 2 puffs until at day six 10 puffs are reached. At day seven 1 puff of Staloral Birch 300 I.R./ml is taken, at day eight 2 puffs and day nine 4 puffs. From then on 4 puffs daily are taken.
  Route of administration: Sublingual application. Drops (for SUBLIVAC Birch) or puffs (for Staloral Birch) are to be held underneath the tongue and then will be swallowed.
  Duration of treatment: 16-20 weeks per subject (at least 12 weeks for subjects with hazel or alder allergy).

SUMMARY:
Objective of the study is to show, on an exploratory basis, that treatment with SUBLIVAC Birch is also effective compared to treatment with Staloral Birch by means of reduction in allergic symptoms during nasal provocation in subjects suffering from IgE mediated allergic complaints triggered by birch pollen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with allergic rhinoconjunctivitis with or without mild asthma (FEV1 ≥ 70%) due to birch pollen for at least 2 years.
* Use of anti-allergy symptomatic medication in the last birch pollen season (in case of a season with low pollen counts, in one of the two previous years).
* No seasonal allergic complaints induced by birch, grasses or mugwort pollen for at least 4 weeks in the absence of rescue medication during at least the last 2 weeks before the baseline.
* A positive SPT (diameter ≥3 mm) for birch pollen and a positive specific serum anti birch IgE-test (>1 U/ml).
* A positive TNPT with a birch allergen extract containing a concentration of 10, 100 or 1000 AU/ml at the baseline visit.
* Age 18 years and older.
* Subjects shall give a written informed consent.

Exclusion Criteria:

* A positive SPT (diameter ≥ 3mm) for hazel or alder and the maintenance dose will not be reached before 8 October 2009.
* A positive SPT (diameter ≥ 3mm) for pets and symptoms related to concomitant sensitization to pets while having these animals at home.
* A positive SPT (diameter ≥ 3mm) for house dust mite or moulds and clinically relevant symptoms related to concomitant sensitization to house dust mite or moulds, based on the investigator's research (TNPT for example).
* Allergy to any of the excipients of SUBLIVAC Birch or Staloral Birch.
* Chronic asthma or emphysema, particularly with an FEV1 < 70 % of predicted value or use of inhalation corticosteroids outside grass and tree pollen season for more than two episodes and/or longer than fourteen days.
* Specific findings for nose and mouth at screening or rhinoscopy before TNPT.
* Serious immuno-pathological diseases or malignancies (including auto-immune diseases, tuberculosis, HIV).
* Inflammation or infection of the target organ (nose, eyes and lungs).
* Severe atopic dermatitis requiring systemic immuno-suppressive medication.
* Allergen specific immunotherapy treatment for a period longer than 3 months within the last 5 years.
* History of life threatening anaphylactic events, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis.
* A positive pregnancy test, lactation or inadequate contraceptive measures. (adequate measures: oral contraceptives, IUD, condom use and having no sexual relationship with a man)
* Alcohol- or drug abuse.
* Lack of co-operation or severe psychological disorders.
* Completed or ongoing long-term treatment with tranquilizer or psycho active drugs.
* Low compliance or inability to understand instructions/study documents
* Completed or ongoing treatment with anti-IgE-antibody
* Patients being in any relationship or dependence with the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Difference in change of the titrated nasal provocation test (TNPT) between the two treatment groups | 16-20 weeks of treatment

SECONDARY OUTCOMES:
Immunoglobulins, changes in TNPT derived variables | 16-20 weeks of treatment
Determination of specific IgE and specific IgG to birch at the baseline and the end of study. It is expected that changes in specific IgE and IgG will be equal in both treatment groups | 16-20 weeks of treatment
At the baseline and the end of study visit the subject will be asked questions for the evaluation of oral allergy syndrome. It is expected that the reduction of oral allergy syndrome complaints will be equal in both treatment groups. | 16-20 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Klimek, PhD, Study Chair — Zentrum für Rhinologie & Allergologie D-Wiesbaden; Oliver Pfaar, MD, Principal Investigator — Zentrum für Rhinologie & Allergologie D-Wiesbaden
Locations (1):
- Zentrum für Rhinologie & Allergologie, Wiesbaden, Hesse, Germany